CLINICAL TRIAL: NCT06397222
Title: Sintilimab, Bevacizumab Plus Y-90 Selective Internal Radiation Therapy for Patients With Unresectable Intermediate-advanced Hepatocellular Carcinoma: a Prospective, Single-center, Single Arm Trial
Brief Title: Sintilimab Plus Bevacizumab and SIRT for Intermediate-advanced HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-16
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Sintilimab; Bevacizumab; Yttrium-90
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sin-Bev-SIRT (Experimental): Sintilimab, Bevacizumab plus SIRT
  Interventions: Drug: Sin-Bev-SIRT

INTERVENTIONS:
Drug: Sin-Bev-SIRT — Sintilimab 200mg I.V. q3w and bevacizumab 7.5mg/kg I.V. q3w will be started at 3-7 days after the first SIRT. Treatment of sintilimab and bevacizumab will last up to 24 months. Patients will be allowed to have sintilimab or bevacizumab as a sigle agent and will be still considered on study when the other drug cause intolerable toxicity.

SUMMARY:
This study is conducted to evaluate the efficacy and safety of sintilimab, bevacizumab plus Y-90 selective internal radiation therapy (SIRT) for patients with unresectable intermediate-advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a single-center, prospective study to evaluate the efficacy and safety of sintilimab, bevacizumab plus SIRT (Sin-Bev-SIRT) in patient with unresectable HCC.

23 patients with unresectable intermediate-advanced HCC (BCLC B/C stage) will be enrolled in this study. The patients will receive sintilimab (200mg I.V. Q3W) and bevacizumab (7.5mg/kg I.V. Q3W) at 3-7 days after SIRT. Sintilimab and bevacizumab will last up to 24 months, or until disease progresses, intolerable toxicity, withdrawal of informed consent, loss of follow-up, death, or other circumstances that require termination of treatment, whichever occurs first.

The primary end point of this study is Progression free survival (PFS) per mRECIST. The secondary endpoints are PFS per RECIST 1.1, objective response rate (ORR), disease control rate (DCR), overall survival (OS) and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC (BCLC stage B/C or CNLC II/III) with diagnosis confirmed by histology/cytology or clinically
* At least one measurable untreated lesion
* Intrahepatic tumors can be treated with 1-2 sessions of SIRT
* Child-Pugh score 5-7
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Life expectancy of at least 3 months
* Patients with active hepatitis B are allowed, but they need to receive antiviral treatment to achieve a HBV DNA<10^3 IU/mL
* Patients with hepatitis C need to finish the anti-HCV treatment

Exclusion Criteria:

* tumor extent ≥70% liver occupation
* Tumor thrombus involving main portal vein or both the first left and right branches of portal vein
* Vena cava invasion
* Central nervous system metastasis
* Metastatic disease that involves major airways or blood vessels
* Patients who previously received hepatic arterial infusion chemotherapy (HAIC), transarterial chemoembolization (TACE), transarterial embolization (TAE), radiotherapy, systemic therapy for HCC
* History of organ and cell transplantation
* Prior esophageal and/or gastric varices bleeding
* Hepatic dysfunction, such as ascites, esophagogastric varices, hepatic encephalopathy
* Evidence of portal hypertension with high risk of bleeding
* Use of immunosuppressive medications within 4 weeks prior to the first dose of study treatment
* Major surgical procedure or unhealed wound, ulcer, or fracture within 4 weeks prior to the first dose of study treatment
* Any life-threatening bleeding event within the previous 3 months, including the need for blood transfusion, surgical or localized treatment, or ongoing drug therapy
* Peripheral blood white blood cell count <3×10^9/L and platelet count <50×10^9/L
* Prolonged prothrombin time >4 seconds
* Severe organ (heart, lung, kidney) dysfunction
* History of other malignancies
* Co-infection with hepatitis B and C viruses
* Human immunodeficiency virus infection
* Pregnant or lactating patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) according to mRECIST | 3 years
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression free survival (PFS) according to RECIST 1.1 | 3 years
  The time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Objective response rate (ORR) | 3 years
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR) according to mRECIST and RECIST 1.1
Disease control rate (DCR) | 3 years
  The percentage of patients who had a tumor response rating of CR, PR, or stable disease (SD) according to mRECIST and RECIST 1.1
Overall survival (OS) | 3 years
  The time from initiation of treatment until the date of death from any cause.
Adverse Events (AEs) | 3 years
  Number of patients with AEs assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided